CLINICAL TRIAL: NCT05374603
Title: Savolitinib Combine With Durvalumab in Chinese EGFR Wild-type Locally Advanced or Metastatic NSCLC Patients With MET Alteration: An Open-label, Interventional, Multiple-center, Exploratory Trial (SOUND)
Brief Title: Savolitinib Combine With Durvalumab in EGFR Wild-type Locally Advanced or Metastatic NSCLC
Acronym: SOUND
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5083C00002
Record Dates: First submitted 2022-04-29; First posted 2022-05-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Savolitinib combine with Durvalumab (Experimental): single-arm
  Interventions: Drug: Savolitinib; Drug: Durvalumab

INTERVENTIONS:
Drug: Savolitinib — Savolitinib combine with Durvalumab
Drug: Durvalumab — savolitinib plus durvalumab

SUMMARY:
This is an open-label, interventional, multiple-center, exploratory Phase II study sponsored by AstraZeneca Investment(China)Co., LTD. to evaluate the efficacy and safety of Savolitinib combine with Durvalumab in Chinese EGFR wild-type locally advanced or metastatic NSCLC patients with MET alteration.

DETAILED DESCRIPTION:
Successfully enrolled, eligible patients will receive treatment of durvalumab (1500 mg, ivgtt, q4w) in combination with savolitinib (600mg for BW≥50kg, 400mg for BW<50kg, p.o., q.d.) after informed consent signed. Treatment will continue until either objective disease progression, unacceptable toxicity occurs, consent is withdrawn, other discontinuation criterion is met, or study completion.

Tumor assessment is conducted according to RECIST 1.1. Baseline tumor assessments should include CT/MRI of chest and abdomen (including liver and adrenal glands) and should be performed within 28 days prior to receiving first dose of treatment. Follow-up assessments should be performed every 8 weeks (±7 days) after the start of treatment until 4 month, and then every 12 weeks until objective disease progression as defined by RECIST 1.1 even if a patient discontinues treatment prior to progression (unless they withdraw consent). Patients who have been observed CR or PR firstly will be scheduled for an additional visit to confirm efficacy at 4 weeks (+7 days) after the first assessment result of CR or PR was observed.

Safety information should be visit in siteand will be prospectively collected from informed consent to the end of the follow-up period, defined as 3028 days (± 7 days) after last dose of Savolitinib, or 90 days (± 7 days) after last dose of Durvalumab which comes later.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses.
3. Females and/or males age ≥18 years at the time of signing the ICF.
4. Body weight >30 kg
5. NSCLC with the following features:

   1. Histologically or cytologically confirmed locally advanced or metastatic NSCLC
   2. EGFR wild-type
   3. MET Exon 14 skipping mutation, or MET overexpression (IHC 3+ in ≥70% of tumor cells), or MET amplification based on FISH (GCN≥5 or MET/CEP7≥2) or NGS (≥20% tumor cells, coverage of ≥200 × sequencing depth and ≥5 copies of MET over tumor ploidy)
6. WHO/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing
7. A minimum life expectancy of 12 weeks at the time of signing the ICF.
8. Patients must have received no more than 2 system anti-cancer treatment at the time of signing the ICF.
9. Patients must have measurable disease per RECIST 1.1, as defined by at least 1 lesion that can be accurately measured at baseline as ≥10 mm at the longest diameter (except lymph nodes which must have a short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI), which is suitable for accurate repeated measurements.
10. Adequate haematological function defined as:

    1. Haemoglobin ≥9 g/dL (no transfusion in the past 2 weeks).
    2. Absolute neutrophil count ≥1.5×109/L.
    3. Platelet count ≥100,000/μL (no transfusion in the past 10 days)
11. Adequate liver function defined as:

    1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x the upper limit of normal (ULN) with total bilirubin TBL ≤1 x ULN
    2. OR TBL >1 x ULN to ≤1.5x ULN with ALT and AST ≤ 1 x ULN
12. Adequate renal function defined as a serum creatinine <1.5 times the institutional ULN OR a glomerular filtration rate ≥50 mL/min, as assessed using the standard methodology at the investigating centre (eg, Cockcroft-Gault, Modification of Diet in Renal Disease or Chronic Kidney Disease Epidemiology Collaboration formulae, ethylenediaminetetraacetic acid clearance or 24-hour urine collection). Confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
13. Adequate coagulation parameters, defined as: International Normalisation Ratio (INR) <1.2 x ULN and activated partial thromboplastin time (aPTT) <1.2 x ULN unless patients are receiving therapeutic anticoagulation which affects these parameters
14. Patients with known tumour thrombus or deep vein thrombosis are eligible if clinically stable on low molecular weight heparin (LMWH) for ≥2 weeks.
15. Ability to swallow and retain oral medications.
16. Willingness and ability to comply with study and follow-up procedures.
17. Females of childbearing potential should be willing to use adequate contraceptive measures (see Section 5.3.1), should not be breast feeding, and must have a negative pregnancy test if of childbearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

    Post-menopausal is defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments; women under the age of 50 years would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution; or women with documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

    Further information is available in Appendix G (Contraception Requirements).
18. Male patients with a female partner of childbearing potential should be willing to use barrier contraception during the study and for 6 months following discontinuation of study drug. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing study treatment.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. As judged by the investigator, active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhoea Grade≥2, malabsorption syndrome or previous significant bowel resection). therapy (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhoea Grade

   ≥2, malabsorption syndrome or previous significant bowel resection).
2. Any of the following cardiac diseases diagnosed currently or within the last 6 months:

   1. Unstable angina pectoris
   2. Congestive heart failure (New York Heart Association [NYHA] ≥Grade 2)
   3. Acute myocardial infarction
   4. Stroke or transient ischemic attack
   5. Ventricular arrhythmias
3. Uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) ≤28 days of beginning study drug.
4. Mean resting correct QT interval (QTcF) >470 msec for women and >450 msec for men at Screening, obtained from 3 ECGs using the screening clinic ECG machine derived QTcF value.

   (a)Any factors that may increase the risk of QTcF prolongation or risk of arrhythmic events such as heart failure, chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes.
5. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECGs ≤28 days of beginning study drug, eg, complete left bundle branch block, third degree heart block, second degree heart block, P-R interval >250 msec.
6. Acute coronary syndrome diagnosed currently or within the last 6 months.
7. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
8. Major surgical procedures ≤28 days of beginning study drug or minor surgical procedures ≤7 days.
9. Active hepatitis B (HBV) (positive HBV surface antigen [HBsAg] result) or hepatitis C (HCV). Viral testing is not required for assessment of eligibility for the study. Patients with a past or resolved HBV or HCV infection are eligible if:

   1. Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc] or
   2. Positive for HBsAg, but for >6 months have had normal transaminases and HBV DNA levels between 0 to 2000 IU/mL (inactive carrier state) and willing to start and maintain antiviral treatment for at least the duration of the study.
   3. Patients with a past or resolved HBV infection must have monthly monitoring of ALT and HBV DNA
   4. HBV DNA levels >2000 IU/mL but on prophylactic antiviral treatment for the past 3 months and must maintain the antiviral treatment during the study.

   Patients with positive HCV antibody are eligible only if the polymerase chain reaction is negative for HCV ribonucleic acid.
10. History of liver cirrhosis of any origin and clinical stage; or history of other serious liver disease or chronic disease with relevant liver involvement, with or without normal LFTs*, such as

    * Hemochromatosis
    * Alpha-1 Antitrypsin deficiency
    * Autoimmune hepatitis (AIH)
    * Primary sclerosing cholangitis (PSC)
    * Primary biliary cirrhosis (PBC)
    * Biopsy-confirmed Non-Alcoholic Steatohepatitis (NASH) with advanced fibrosis
    * Biopsy- confirmed Alcoholic Steatohepatitis with advanced fibrosis
    * Wilson's disease.
    * Hepatocellular carcinoma* Patients with liver metastases are eligible, provided they meet other eligibility criteria, including liver biochemistry criteria.
11. Presence of other active cancers, or history of treatment for invasive cancer, within the last 5 years. Patients with Stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (ie, non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
12. Having gene mutations sensitive to targeted drugs for EGFR, ALK and ROS-1.
13. Unresolved toxicities from any prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment with the exception of alopecia
14. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study intervention. Subjects with leptomeningeal metastases are ineligible.
15. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
16. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc].

    The following are exceptions to this criterion:
    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the Study Physician
    5. Patients with celiac disease controlled by diet alone
17. Known serious active infection including, but not limited to, tuberculosis, or human immunodeficiency virus (positive human immunodeficiency virus 1/2 antibodies). Testing is not required for assessment of eligibility for the study.
18. Known contraindications to durvalumab administration.
19. Known hypersensitivity to the active or inactive excipients of durvalumab or savolitinib or drugs with a similar chemical structure or class.
20. Prior exposure to immune-mediated therapy including, but not limited to, other anti CTLA-4, anti-PD-1, anti-PD-L1, and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, excluding therapeutic anticancer vaccines.
21. Prior exposure to any HGF/MET inhibitor, e.g., foretinib, crizotinib, cabozantinib, merestinib, onartuzumab, capmatinib, tepotinib, etc.
22. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including renal transplant, active bleeding diatheses or uncontrolled hypertension, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol.
23. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, targeted therapy, biologic therapy, tumor embolisation, or monoclonal antibodies) of early stage NSCLC within 14 days prior to the first dose of study intervention.
24. Participation in another clinical study with a study intervention or investigational medicinal device administered in the last 30 days prior to the first dose of study intervention or concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the off-treatment follow-up period of an interventional study.
25. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
26. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
27. Previous enrolment in the present study.
28. Without civil capacity or with restricted civil capacity.
29. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
30. Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab. Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab
31. Any other reasons judged by the leading investigator to prevent the subject from participating in this study
32. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4, strong inhibitors of CYP1A2, within 2 weeks of the first dose of study treatment (3 weeks for St John's Wort) will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
PFS | The analysis will occur when 60 percent PFS event is observed in each cohort, at approximately 10 months after last patient in.
  PFS (Progression-Free Survival ) will be defined as the time from first dose of study intervention until progression per RECIST 1.1 as assessed by the investigator or death due to any cause prior to progressive disease.

SECONDARY OUTCOMES:
ORR | The analysis will occur at two months after last patient in.
  ORR(Objective Response Rate) defined as the proportion of participants who achieved a CR (Complete Response) or PR(Partial response) as their best overall response based on Response Evaluation Criteria in Solid Tumors (RECIST)1.1 as assessed by the investigator.
DoR | The analysis will occur when 60 percent PFS event is observed in each cohort, at approximately 10 months after last patient in.
  DoR(Duration of Response)is defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression (ie, date of PFS (Progression-Free Survival ) event or censoring-date of first response+1).
DCR | The analysis will occur at two months after last patient in.
  DCR (Disease Control Rate)is defined as the number(percent)of subjects with at least one visit response of confirmed CR (Complete Response), PR (Partial Response) or SD(Stable Disease), based on based on Investigator assessment according to RECIST 1.1.
OS | The analysis will occur when 60 percent PFS event ratio is observed in each cohort, at approximately 10 months after last subject in, up to a maximum of approximately 3 years after first subject in.
  OS(Overall Survival) is defined as the time from the start of treatment until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.

OTHER OUTCOMES:
PD-L1 expression | The analysis will occur at two months after last patient in.
  To explore the efficacy of savolitinib plus durvalumab across different PD-L1 expression level.
Gene profile | The analysis will occur when 60 percent PFS event is observed in each cohort.
  To assess the gene profile in Chinses patients with MET alteration.
Potential molecular resistance mechanism | The analysis will occur when 60 percent PFS event is observed in each cohort.
  To explore potential molecular resistance mechanism at disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Doctor, Principal Investigator — Shanghai Chest Hospital
Locations (12):
- China (12):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chongqing
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trails via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrails.pharmacm.com/ST/Submission/Disclosure.
  Indicates that AZ accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrails.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in approved sponsored tool. Signed Data Sharing Agreement(non-negotiable contract for data accessors)must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MES to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrails.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home